CLINICAL TRIAL: NCT01391208
Title: A Phase I In-Vivo Esophageal Protocol for Detection of Neoplasia in the Digestive Tract
Brief Title: Esophageal Protocol for Detection of Neoplasia in the Digestive Tract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Missy Tuck, Project manager, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U54CA136429 (NIH)
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett's Esophagus with High Grade Dysplasia; Esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peptide application (No Intervention)
  Interventions: Drug: GI heptapeptide

INTERVENTIONS:
Drug: GI heptapeptide — GI heptapeptide, Linear, 7 amino acid peptide sequence ASYNYDA with a 5-FITC tag and NH2 terminus. Chemical Formula: Ala1-Ser2-Tyr3-Asn4-Tyr5-Asp6-Ala7-Gly8- Gly9-Gly10-Ser11-Lys12 (5-FITC) -NH213.Investigational Agent Manufacturer: CPC Scientific, 1245 Reamwood Ave, Sunnyvale, CA 94089 Investigational Agent information: Lot Number: 10031701, M.W. 1577.6, 97.2% pure. Stored at -20C Yellow, lyophilized powder in single use amber vials. 5-FITC is light-sensitive, therefore stored protected from light. Manufactured under cGMP with Certificate of Analysis (COA) provided.

SUMMARY:
You are invited to participate in a research study to develop new ways to look for abnormal areas/tissues of the esophagus. The current endoscopes used to look at the esophagus are very good, but if the area doesn't look different to the naked eye, then the endoscope can't improve on that. The investigators are looking at using special fluorescent stains in addition to special endoscopes designed to see abnormal areas that are not obvious to the naked eye. Currently specialized microscopes and fluorescent stains are used in clinical laboratories but it takes several days of processing to get results. It may be very helpful to look for areas to sample for abnormal tissue during the endoscopy procedure.

You are being asked to let us use "fluorescent peptides" with a special endoscope that allow us to "see" of your esophagus with both fluorescent and white light during your upper GI endoscopy procedure to help target your biopsies. Peptides are small chains of amino acids (the building blocks that make up proteins) linked together. Our peptide is a chain of 7 amino acids attached to a fluorescent dye called FITC (like the one used by your eye doctor).

The investigators have prepared special "fluorescent peptides", that will "glow" when a special light is used that should help us separate normal tissue from abnormal tissue. In this study, the investigators will apply the special fluorescent peptides by a spray catheter to your esophagus to help us target you biopsies. Both routine and targeted biopsies will be taken as your endoscopist feels is indicated.

This is a phase 1 study. This means that this is the first time the investigators have used this kind of "fluorescent peptide" in people. The Food and Drug Administration (FDA) has not approved this agent, but is allowing us to test it in this study. The main goal of this study is to see if there are any side effects from using the peptide. Our second goal is to see if the peptide "glows" well and if the investigators can take pictures of the areas that do glow.

This is the first test of this agent, so it won't be used to change how your biopsies are taken nor how your endoscopy is done.

DETAILED DESCRIPTION:
SUMMARY OF STUDY PLAN A Phase I study of the safety of a topically-administered 7-amino acid peptide with a fluorescein analog (5-FITC) label for detecting neoplastic areas of the esophagus is proposed. The study will test the safety of administering this agent (5-FITC-labeled 7-AA peptide) to human subjects undergoing clinically-indicated upper endoscopy and/or endoscopic ultrasound for suspected esophageal adenocarcinoma with or without Barrett's Esophagus or High-Grade dysplasia (HGD) in Barrett's Esophagus. We intend to enroll 25 evaluable subjects. We expect to be able to enroll about 5 subjects per month, so the study should take about 6-9 months to complete.

Subjects will be recruited around their scheduled procedure. The endoscopists performing the procedures are all investigators on this protocol and on the FDA form 1572. Blood for clinical labs and urine for dipstick urinanalysis (and pregnancy test, if applicable) will be collected pre-procedure, along with medical information. Vital signs are monitored throughout the clinical procedure and will be captured on case report forms, so no separate physical exam is necessary. The endoscopy will proceed per UMHS (University of Michigan Health System) standard of care and guidelines for management of Barrett's Esophagus (American College of Gastroenterology, Appendix C). The endoscopist performing the clinical procedure will evaluate the potential risk (if any) for their patient to continue with the procedure or study. The endoscopist will spray the reconstituted 5-FITC-labeled peptide onto the esophageal mucosa through a catheter in the endoscope. Pictures with white-light will be taken with the standard endoscope before and after the peptide application. The Mauna Kea/Cellvizio® or miniprobe , an FDA approved instrument (510(k) ref # K051585) will be passed through the instrument channel of the standard endoscope and used for collecting confocal images of up to two areas where the peptide binds. Biopsies will taken as clinically indicated, including the two places where the confocal images were taken. Data about all clinical biopsies will be collected on case report forms. All biopsies are for clinical care only (not research use) and will be sent for routine histology per UMHS standard of care.

Approximately 24 hours (± 4 hours) post-procedure, blood for clinical labs and urine for dipstick urinanalysis (UA) will be collected to assess for potential effects (if any) from applying the peptide solution. Subjects will receive compensation for the inconvenience of returning for another blood draw. Subjects may be able to have their blood and UA done at a UMHS lab or QUEST Diagnostics Lab closer to their home Subjects will receive compensation for the inconvenience of returning for another blood draw. Subjects may be able to have their blood and UA done at a UMHS lab or QUEST Diagnostics Lab closer to their home orby Michigan Clinical Research Unit to you (MCRU 2U). Additional blood draws for follow up labs may be needed if any significant differences from baseline are seen. Additional compensation will be offered for those blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have biopsy-proven or suspected high-grade dysplasia or esophageal adenocarcinoma with or without confirmed Barrett's Esophagus.
* Subjects who are scheduled for a clinically-indicated upper endoscopic evaluation and/or intervention (e.g. esophagogastroduodenoscopy (EGD) with biopsies).
* All subjects who are medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities) who meet the inclusion/exclusion will be included. Standard practice guidelines for safely proceeding with the procedure will be sufficient for our study.
* Adults aged 18 years to 100 years old.
* Willing and able to sign informed consent.
* The effects of the 5-FITC-labeled peptide on the developing human fetus are unknown. For this reason, women of child-bearing potential must have a negative pregnancy test on the day of the procedure to receiving the 5-FITC-labeled peptide agent or be post-menopausal. Post-menopausal women are defined as post-hysterectomy, or over 40 and at least 18 months without menses and not on birth-control.

Exclusion Criteria:

* Subjects with known allergy or negative reaction to fluorescein or derivatives.
* Subjects who have had an esophagectomy.
* Subjects who are also prepped for colonoscopy with the EGD.
* Subjects on active chemotherapy or radiation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety of peptide application | 0 (baseline) and 24 hours
  The study will test the safety of administering this agent to human subjects. Prior to the EGD,subjects will have baseline blood work, urinanalysis via dipstick and urine pregnancy test. Labs for CBC w/ platets, chemistries and liver function tests and (COMP panel). These labs will be to compare to post-procedure levels for any possible side effects. These tests will be repeated 24 hours post peptide application and as needed weekly until labs resolve to normal ranges.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States